CLINICAL TRIAL: NCT06484582
Title: Investigation of Musculoskeletal System Disorders Seen in Automotive Industry Workers
Status: Recruiting | Type: Observational
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Other Study IDs: Uskudar13
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Work-related Illness; Work Injury
MeSH Terms: interventions — Workforce

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: workers — This study will be conducted as a face-to-face survey. Surveys will be created with Google Forms and will be filled out by the physiotherapist according to the participant's response.

SUMMARY:
The aim of this study is to examine the musculoskeletal disorders seen in automotive industry workers.

DETAILED DESCRIPTION:
This study will be conducted as a face-to-face survey. Surveys will be created with Google Forms and will be filled out by the physiotherapist according to the participant's response.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 25-60
* Not having any psychological or neurological disorders
* Being able to communicate in Turkish (written, verbal)
* Being able to communicate cognitively adequately
* Working full-time
* Being employed in an automotive industry for at least 5 years

Exclusion Criteria:

* Being under 18 or over 60
* Working part-time
* Being employed in the same business for less than 5 years

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: auto industry workers
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Work Productivity & Activity Impairment Questionnaire - General Health | 1 week
  It is a tool developed to assess how health problems affect working life and daily activities in the general population. It measures the impact of health and symptom severity based on work productivity and leave time assessments and consists of 6 questions. These are; employment status, working hours, hours missed due to health problems, hours missed due to other reasons and the last two questions are the hours actually worked. It is scored from 0 to 10 points. The highest is 70, the lowest is 0. Higher scores indicate prolonged sick leave or impairment and reduced productivity.
Pittsburgh Sleep Quality Survey | 1 week
  The scale includes a total of 24 questions. 19 of these questions are self-evaluation questions, and 5 of them are answered by the individual's spouse or a roommate. These 5 questions are used for clinical information only and are not included in the scoring. The scale questions that determine sleep quality include various factors related to sleep quality. These questions are to determine sleep duration, sleep latency, and the frequency and severity of specific sleep-related problems; 18 items were grouped as 7 component scores. The total score ranges from 0 to 21. A high total score indicates poor sleep quality. The scale does not indicate the presence of sleep disorders or the prevalence of sleep disorders. However, it is stated that a total score of 5 and above indicates poor sleep quality.
Disabilities of the Arm, Shoulder and Hand Questionnaire | 1 week
  It was developed to evaluate functional status and symptoms by focusing on physical function in upper extremity injuries. According to the results of the survey; a result from 0-100 is obtained from each part; 0-no apology 100-maximum apology.
Rapid Upper Limb Assessment | 1 week
  It is an ergonomics risk assessment method that quickly analyzes the employee's upper extremity from an ergonomic perspective. It evaluates upper extremity movements in 14 separate steps. 8 of these steps are scored for arm and hand position, and 6 for neck and trunk position, according to the table. The minimum Rapid Upper Limb Assessment Score = 1, and the maximum Rapid Upper Limb Assessment Score = 7. A high score means high risk.
Nordic Extended Musculoskeletal Questionnaire | 1 week
  It is one of the questionnaires used to evaluate the severity and impact of musculoskeletal symptoms. In the survey, the frequency and severity of pain in the 'Neck, Shoulder, Upper Back, Elbow, Hand-wrist, Kala, Knee, Foot-ankle' areas of the body are evaluated in the last 12 months.It is a selection scale rather than a rating.
The McGill Pain Questionnaire | 1 week
  McGill pain questionnaire-short form is used to evaluate patients' pain in terms of feeling and sensory. Pain level is defined with 15 words consisting of 11 sensory and 4 affective words. From these descriptive words, the patient should choose an answer that is compatible with him/her as "no (0)", "mild (1)", "moderate (2)", "severe (3)". In addition, the pain felt during the survey is measured with the Visual analog scale , and the total pain intensity of the pain is measured with a 6-point Likert scale. Pain is defined as "absent (0)" and "unbearable (5)" on the Likert scale. In total, pain scores between 0-45 (no pain=0, severe pain=45).

CONTACTS AND LOCATIONS:
Overall Officials: Sude Asya ALŞAN, Study Chair — Uskudar University
Locations (1):
- Uskudar University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eakin JM. Leaving it up to the workers: sociological perspective on the management of health and safety in small workplaces. Int J Health Serv. 1992;22(4):689-704. doi: 10.2190/DNV0-57VV-FJ7K-8KU5. PMID 1399176
- [Background] Govaerts R, Tassignon B, Ghillebert J, Serrien B, De Bock S, Ampe T, El Makrini I, Vanderborght B, Meeusen R, De Pauw K. Prevalence and incidence of work-related musculoskeletal disorders in secondary industries of 21st century Europe: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2021 Aug 31;22(1):751. doi: 10.1186/s12891-021-04615-9. PMID 34465326
- [Background] d'Errico A, Cardano M, Landriscina T, Marinacci C, Pasian S, Petrelli A, Costa G. Workplace stress and prescription of antidepressant medications: a prospective study on a sample of Italian workers. Int Arch Occup Environ Health. 2011 Apr;84(4):413-24. doi: 10.1007/s00420-010-0586-3. Epub 2010 Oct 16. PMID 20953623
- [Background] da Costa BR, Vieira ER. Risk factors for work-related musculoskeletal disorders: A systematic review of recent longitudinal studies. Am J Ind Med. 2010 Mar;53(3):285-323. doi: 10.1002/ajim.20750. PMID 19753591